CLINICAL TRIAL: NCT03177031
Title: A Randomised, Open-label, Parallel Group, Multi-centre Controlled Study to Evaluate the Clinical Performance and Safety of Stay Safe Link® Compared With Stay Safe® in Patients With End-stage Kidney Disease on Continuous Ambulatory Peritoneal Dialysis
Brief Title: Clinical Performance and Safety Comparison of Stay Safe Link® With Stay Safe® in Patient on CAPD (CAPD-3)
Acronym: CAPD-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HPP/CTP/PD/003
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Continuous Ambulatory Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stay Safe (STS) (Active Comparator): CAPD system produced by Fresenius Medical Care in Germany
  Interventions: Device: Stay Safe (STS)
- Stay Safe Link (SSL) (Experimental): CAPD system produced by Fresenius Medical Care in Malaysia
  Interventions: Device: Stay Safe Link (SSL)

INTERVENTIONS:
Device: Stay Safe Link (SSL) — CAPD system produced in Malaysia by Fresenius Medical Care
  Arms: Stay Safe Link (SSL)
Device: Stay Safe (STS) — CAPD system produce in Germany by Fresenius Medical Care
  Arms: Stay Safe (STS)

SUMMARY:
This post-marketing study is undertaken to compare the clinical effectiveness and safety of two continuous ambulatory peritoneal dialysis produced by Fresenius Medical Care (FMC), i.e. Stay Safe® (STS) that is produced by a plant in Germany and Stay Safe Link® (SSL) that is produced in Malaysia. The study is an open labelled, randomised controlled trial where 434 patients in total will be randomised to either STS or SSL in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or above
2. End stage kidney failure receiving Stay Safe® PD system for at least 4 weeks
3. Written informed consent

Exclusion Criteria:

1. Requirement for 2.5L exchanges
2. Requirement for Stay Safe Balance®
3. PD-related infection (peritonitis, exit site or tunnel tract infection) in the preceding 8 weeks or during conversion
4. Malfunctioning of PD catheter
5. Planned transfer to automated peritoneal dialysis, haemodialysis or transplant within 90 days
6. Pregnancy
7. Any condition that compromises the integrity of the abdominal wall, abdominal surface, or intra-abdominal cavity, such as documented loss of peritoneal function
8. History of active alcohol or substance abuse in the previous 6 months
9. Other medical condition which, in the investigator's judgement, may be associated with increased risk to the subject or may interfere with study assessments or outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Peritonitis Rate of Stay Safe Link system | 1 year

SECONDARY OUTCOMES:
Dialysis dose delivered | 1 year
  weekly Kt/V
Dialysis dose delivered | 1 year
  creatinine clearance (L)
Ultrafiltration volume | 1 year
  Post-PD bodyweight (kg) minus Pre-PD bodyweight (kg)
Product deficiencies of the PD system | 1 year
  Defect or leakages of PD bags, tubing or organiser (number of defects or leakages detected)
Product deficiencies of the PD system | 1 year
  Bacterial or other contamination of dialysate or any component of the PD system (number of contamination detected)
Safety Assessment of the PD system | 1 year
  Technique failure, defined as the transfer to hemodialysis for more than 30 days (number of technique failure detected)

CONTACTS AND LOCATIONS:
Overall Officials: Loke Meng Ong, Principal Investigator — Clinical Research Centre, Penang General Hospital, Malaysia
Locations (1):
- Clinical Research Centre, Penang Hospital, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers

REFERENCES:
- [Derived] Mak WY, Ong LM, Goh BL, Bavanandan S, Mushahar L, Leong CT, Hooi LS. Protocol for a randomised, open-label, parallel group, multicentre controlled study to evaluate the clinical performance and safety of Stay Safe Link compared with Stay Safe in patients with end-stage kidney disease on continuous ambulatory peritoneal dialysis. BMJ Open. 2019 Mar 8;9(3):e024589. doi: 10.1136/bmjopen-2018-024589. PMID 30852538